CLINICAL TRIAL: NCT02304237
Title: A Multicenter, Randomized, Open-label, Investigator Initiated Trial of Vaginal Compared With Intramuscular Progesterone for Prevention of Preterm Birth in High Risk Pregnant Women
Brief Title: Vaginal Compared With Intramuscular Progesterone for Prevention of Preterm Birth in High Risk Pregnant Women
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Collaborators: Samsung Medical Center (Other); Han Wha Pharma Co., Ltd. (Industry); Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Young Ju Kim, Professor, Ewha Womans University Mokdong Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VICTORIA
Record Dates: First submitted 2014-11-26; First posted 2014-12-01 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Premature Birth
Keywords: Premature Birth; progesterone
MeSH Terms: conditions — Premature Birth | interventions — Utrogestan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal progesterone (Experimental): Vaginal progesterone(Utrogestan)200mg/day, during 14~21 weeks.
  Interventions: Drug: Vaginal progesterone
- Intramuscular progesterone (Active Comparator): Intramuscular progesterone(Progesterone Depot Jenapharm Injection)250mg/week, during 14~21 weeks.
  Interventions: Drug: Intramuscular progesterone

INTERVENTIONS:
Drug: Vaginal progesterone — micronized progesterone 200mg/day till 36 weeks 6 days of gestation or premature rupture of membranes
  Other Names: Utrogestan
  Arms: Vaginal progesterone
Drug: Intramuscular progesterone — hydroxyprogesterone caproate 250mg/ml/week till 36 weeks 6 days of gestation or premature rupture of membranes
  Other Names: Progesterone Depot Jenapharm Injection
  Arms: Intramuscular progesterone

SUMMARY:
This study is for compare the efficacy of two different regimens(vaginal vs intramuscular) of progesterone therapy in prevention of preterm birth in high risk pregnant women.

DETAILED DESCRIPTION:
The objectives of this study is 1) To compare the efficacy of two different regimens of progesterone therapy in preventing preterm birth less than 37 weeks of gestation. 2) To compare the cost-benefit, adverse effects and patient preference of two different regimens of progesterone therapy.

Design: Multi-center, randomized, open-label trial

ELIGIBILITY:
Inclusion Criteria:

* With a history of prior spontaneous preterm birth or short cervix length
* Spontaneous preterm birth: preterm birth <37 weeks of gestation due to spontaneous preterm labor or preterm premature rupture of membranes (PPROM)
* Short Cervix length : cervix length <25 mm as measured by transvaginal ultrasound at 16-24 weeks of gestation

Exclusion Criteria:

* Multiple gestations
* Major congenital anomalies
* Elective prophylactic cervical cerclage <16 weeks of gestation during current pregnancy
* Previous intentional preterm birth due to maternal or fetal indications, such as preeclampsia and fetal growth restriction
* Diabetes, hypertension, other severe medical diseases

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Preterm Birth Rate before 37 weeks of gestation | from study enrollment to maximum 37 weeks of gestation

SECONDARY OUTCOMES:
Preterm Birth Rate before 34 weeks of gestation | from study enrollment to maximum 34 weeks of gestation
Preterm Birth Rate before 28 weeks of gestation | from study enrollment to maximum 28 weeks of gestation
Result of birth(rate of death, weight, cause of hospitalization to NICU) | from study enrollment to maximum 37 weeks of gestation
Any complications occurred to newborn and mother | from study enrollment to maximum 37 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Young Ju Kim, Principal Investigator — Ewha Womans University Mokdong Hospital

REFERENCES:
- [Derived] Choi SJ, Kwak DW, Kil K, Kim SC, Kwon JY, Kim YH, Na S, Bae JG, Cha HH, Shim JY, Oh KY, Lee KA, Kim SM, Cho IA, Lee SM, Cho GJ, Jo YS, Choi GY, Choi SK, Hur SE, Hwang HS, Kim YJ; from The Preterm Birth Research Committee of the Korean Society of Maternal Fetal Medicine. Vaginal compared with intramuscular progestogen for preventing preterm birth in high-risk pregnant women (VICTORIA study): a multicentre, open-label randomised trial and meta-analysis. BJOG. 2020 Dec;127(13):1646-1654. doi: 10.1111/1471-0528.16365. Epub 2020 Jul 14. PMID 32536019